CLINICAL TRIAL: NCT03379220
Title: Development and Validation of Spreading Depolarization Monitoring for TBI Management
Brief Title: Spreading Depolarizations in Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jed Hartings, Research Associate Professor, University of Cincinnati
Other Study IDs: Hartings SD-II
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Subdural ECoG (Group 1): For patients who require craniotomy to treat TBI, a subdural electrode strip will be placed intraoperatively following evacuation of a hematoma or contusion, as required. Electrode strips will be used for subsequent electrocorticography (ECoG) during intensive care. Patients will also undergo continuous scalp EEG monitoring.
- Burr Hole ECoG (Group 2): For patients who do not require surgery but do require invasive monitoring, an intraparenchymal ECoG electrode array will be placed through a cranial burr hole. Depending on other monitoring needs, the location of injuries, and other clinical considerations, the burr hole may be the same as used for placement of other probes or may be separate. In cases of focal injury, the burr hole will be placed to allow electrode targeting to a lobe with significant primary lesion(s). Patients will also undergo continuous scalp EEG monitoring.
- EEG (Groups 1-3): Continuous EEG recordings will be made using Ag/AgCl electrodes placed on or beneath the scalp (subdermal wire) according to standard practice. The default montage will employ eight lead electrodes for each hemisphere following the 10/20 system (Right: Fp2, F4, C4, P4, O2, F8, T4, T6; left: Fp1, F3, C3, P3, O1, F7, T3, T5). Other montages with more dense placement of electrodes in the region of ECoG monitoring may also be used.

SUMMARY:
This research aims to extend the application of spreading depolarization monitoring to non-surgical TBI patients, using intraparenchymal electrode arrays and scalp electroencephalography to detect depolarizations and develop less invasive monitoring methods.

DETAILED DESCRIPTION:
This study aims to develop the new clinical science of spreading depolarizations for routine monitoring of all TBI patients requiring intensive care. This will be accomplished by investigating automated and non-invasive methods for bedside detection of spreading depolarizations and by determining the prognostic value of such monitoring across the spectrum of TBI severity. While current monitoring of depolarizations is invasive and limited to the subgroup of TBI patients requiring craniotomy, pilot studies have shown that spreading depolarizations are also manifested in non-invasive scalp electroencephalographic (EEG) recordings. Here, approximately 189 subjects will undergo neuromonitoring with EEG only (n=63), with combined EEG and intraparenchymal ECoG (n=63), or with combined EEG and subdural ECoG (n=63). Simultaneous ECoG and EEG monitoring will allow characterization of the EEG signatures of spreading depolarizations and enable identification of signal-processing steps and quantitative criteria for their detection with clinically meaningful sensitivity and specificity, as validated against the gold standard of invasive ECoG. In parallel, an observational electrophysiology study of all TBI patients admitted to intensive care, including non-surgical cases, will characterize the incidence of spreading depolarizations across the TBI severity spectrum. Successful completion of these objectives will 1) determine the extent to which findings obtained in surgical TBI patients also generalize to patients who are managed medically, and 2) establish the first non-invasive method for routine bedside monitoring of a neuronal pathomechanism with proven relevance to TBI outcome. In doing so, this study may enable an individualized approach to TBI management and clinical trials in which neuroprotective therapies can be administered selectively to patients based on real-time identification of a marker and mechanism of secondary neuronal injury.

ELIGIBILITY:
Inclusion Criteria:

1. Enrollment in TRACK-TBI CA cohort
2. Admission to intensive care
3. Documented TBI <24 hr before anticipated placement of electrodes
4. Lobe of primary injury accessible for ECoG by burr hole or craniotomy access
5. Age ≥ 18 years
6. Acute brain CT for clinical care
7. Visual acuity/hearing adequate for testing
8. Fluency in English or Spanish
9. Ability to obtain informed consent

Exclusion Criteria:

1. Significant polytrauma that would confound outcome assessment
2. Prisoners or patients in custody
3. Pregnancy
4. Patients on psychiatric hold
5. Major debilitating baseline mental health disorder that would interfere with follow-up and the validity of outcome
6. Major debilitating neurological disease impairing baseline awareness, cognition, or validity of follow-up and outcome assessment
7. Significant history of pre-existing conditions that would interfere with follow-up and outcome assessment
8. Low likelihood of follow-up
9. Current participation in an interventional trial
10. Penetrating TBI
11. Spinal cord injury with ASIA score of C or worse
12. Bilateral unreactive pupils or other evidence of unsurvivable injury
13. Evidence of coagulopathy (INR>1.5 or thrombocytopenia) or infection, which contraindicate invasive monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 189 patients admitted to intensive care for treatment of TBI will be enrolled. The study will be conducted as an addition to TRACK-TBI (Transforming Research and Clinical Knowledge in Traumatic Brain Injury), an observational study conducted at 11 sites in the United States. The present study will be implemented at 7 of the 11 sites: University of Cincinnati, University of Pennsylvania, University of Pittsburgh, University of Miami, Massachusetts General Hospital, University of California San Francisco, and Baylor College of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended (GOS-E) | 6 months following injury
  Glasgow Outcome Scale- Extended (GOS-E) is an ordinal global scale for functional outcome that rates patient status into one of eight categories, with higher scores representing better recovery: Dead (1), Vegetative State (2), Lower Severe Disability (3), Upper Severe Disability (4), Lower Moderate Disability (5), Upper Moderate Disability (6), Lower Good Recovery (7), and Upper Good Recovery (8).

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas